CLINICAL TRIAL: NCT03896425
Title: Increased Thalamocortical Connectivity in Tdcs-potentiated Generalization of Cognitive Training
Brief Title: Maximizing the Impact of Neuroplasticity Using Transcranial Electrical Stimulation Study 1
Acronym: MINUTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26586_01; 1RF1MH116987-01 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Transcranial Direct Current Stimulation; Healthy
Keywords: tDCS; cognitive training; functional connectivity; non-invasive brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- right active-tDCS (Experimental): 2-3 times/week for 12 weeks: ramp-up for 30 seconds, 2mA right (AF4 anode - AF3 cathode) for 20 min, and then ramp-down for 30 seconds.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- left active-tDCS (Experimental): 2-3 times/week for 12 weeks: ramp-up for 30 seconds, 2mA left (AF3 anode - AF4 cathode) for 20 min, and then ramp-down for 30 seconds.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- sham tDCS (Sham Comparator): Current will be turned off immediately after the initial 30-second ramp-up period.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Three different stimulation montages will be programmed: right, left and sham. During the Ramp periods, 2 mA current will be delivered to both AF3 and AF4 with an ascending (RampUp) and descending ramp (RampDown) over 30 sec via two saline soaked electrode sponges (~ 25cm²; current density = 0.08 mA/cm²). In this way, all subjects experience the same sensation on both sides to blind them to condition. During the Constant period, current will be set based on the Condition: Right - 2mA AF4 anode-AF3 cathode; Left - 2mA applied to AF3 anode-AF4 cathode; Sham - current turned off.

SUMMARY:
Non-invasive neuromodulation, such as transcranial direct current stimulation ( tDCS) , is emerging as an important therapeutic tool with documented effects on brain circuitry, yet little is understood about h ow it changes cognition. In particular, tDCS may have a critical role to play in generalization, that is how training in one domain generalizes to unlearned or unpracticed domains. This problem has resonance for disorders with cognitive deficits, such as schizophrenia.

Understanding how tDCS affects brain circuity is critical to the design and application of effective interventions, especially if the effects are different for healthy vs. psychiatric populations. In previous research, one clue to the mechanism underlying increased learning and generalization with tDCS was provided by neuroimaging data from subjects with schizophrenia undergoing cognitive training where increases in thalamocortical (prefrontal) functional connectivity (FC) predicted greater generalization.

The premise of this proposal is that increases in thalamocortical FC are associated with the generalization of cognitive training, and tDCS facilitates these increases. The overarching goals of this proposal are to deploy neuroimaging and cognitive testing to understand how tDCS with cognitive training affect thalamocortical circuitry in individuals with and without psychosis and to examine variability in response within both groups.

Study 1 will compare right prefrontal, left prefrontal and sham tDCS during concurrent cognitive training over 12 weeks in 90 healthy controls. Study 2 (NCT03896438) will be similar in all aspects but will examine 90 patients with schizophrenia or schizoaffective disorder and include clinical assessments. Results of the study will provide crucial information about location of stimulation, length of treatment, modeled dosage, trajectory and durability needed to guide future research and interventions for cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide consent and comply with study procedures.
2. Age 18 - 60 years old.
3. Estimated IQ range within the range: 70 ≤ IQ ≤ 115.
4. No Serious and Persistent Mental Illness (SPMI) or addictive disorder diagnosis as measured by the MINI (Mini International Neuropsychiatric Interview), or sleep disorder;
5. Ability to participate in three weekly 45' training sessions over 12 weeks and participate in four assessments.

Exclusion Criteria:

1. Any medical condition or treatment with neurological sequelae (e.g. stroke, tumor, loss of consciousness > 30 min, HIV).
2. Contraindications for tDCS or MRI scanning (tDCS contraindication: history of seizures; MRI contraindications: The research team will utilize the CMRR Center's screening tools and adhere to the screening SOP during enrollment of all research participants in this protocol. The CMRR Center's screening tools and SOP are IRB approved under the CMRR Center Grant (HSC# 1406M51205) and information regarding screening procedures is publicly available on the CMRR website (CMRR Policies / Procedures).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Started | 20 | 18 | 20
Completed | 13 | 10 | 15
Not Completed | 7 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 18 | 20 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 20 | 58
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 22.9 (5.3) | 26.6 (8.2) | 24.9 (8.9) | 24.7 (7.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 9 | 6 | 22
  Male | 13 | 8 | 14 | 35
  Nonbinary | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 15 | 15 | 14 | 44
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: Most participants completed MRI sessions on a 3T scanner located in the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota. FC measures how different brain regions change in activation together. We characterized FC using global connectivity from graph theory analysis. We extracted the fMRI time courses from 454 parcellations defined by the 400 S4 Schaefer Atlas (Schaefer et al., 2018) combined with the Melbourne Subcortex Atlas (Tian et al., 2020). We computed the absolute value of the Pearson's correlation for all possible pairs of time series, creating a 454x454 (N x N) connectivity matrix, which was then reduced to 10% most significant connections by subject. We estimated the FC by calculating the node strength for each parcellation, which is the weighted mean of all significant connections, from these connectivity matrices. Finally, we averaged node strength across parcellations to calculate global node strength. Higher values indicate more brain-wide FC.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 18 | 20
arbitrary units | 22.7 (4.0) | 20.5 (4.0) | 21.9 (2.8)

2. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: Task-dependent thalamocortical connectivity associated with the N-back task was calculated by modeling the block task design together with the thalamic regressor using psychophysiological interaction analysis (PPI). The thalamic regressor is the time series of the mediodorsal thalamus from the Melbourne atlas. The primary analysis focused on the 2-back conditions alone. The PPI analysis calculates the functional connectivity between the mediodorsal thalamus and all other brain regions specifically during 2-back trials. Neural activation related to the thalamic regressor was compared to neural activation during the fixation (no choices made) to normalize the relative activation (z-score). Positive values indicate increased functional connectivity with the thalamus during the 2-back choices. A z-score of zero represents no difference compared to the fixation cross (no choices). We report the average z-score of the PPI regressor within the control network (Yeo et al., 2011).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 16 | 20
z-score | -0.58 (0.58) | -0.27 (0.48) | -0.29 (0.34)

3. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: Task-dependent thalamocortical connectivity associated with the Dot Pattern Expectancy (DPX) task demands will be identified by analyzing cue and probe events together with the thalamic regressor using psychophysiological interaction analysis (PPI). The thalamic regressor is the time series of the mediodorsal thalamus from the Melbourne atlas. We examined B-cue related connectivity. The PPI analysis calculates the functional connectivity between the mediodorsal thalamus and all other brain regions specifically during B-cue trials. Neural activation related to the thalamic regressor was compared to neural activation during the fixation (no choices made) to normalize the relative activation (z-score). Positive values indicate increased functional connectivity with the thalamus during the B-cue responses. A z-score of zero represents no difference compared to the fixation cross (no choices). We report the average z-score of the PPI regressor within the control network (Yeo et al., 2011).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 18 | 20
z-score | -0.13 (0.49) | -0.14 (0.32) | -0.18 (0.36)

4. Primary Outcome: D-prime Score
Description: The n-back task measures working memory capacity. The participant is presented with a series of stimuli and instructed to indicate with a button press when the current stimulus matches the stimulus that appeared a pre-determined number (n) of trials before. d' (d prime) will be calculated as a measure of signal detection, which indicates the normalized rate of hits to false positives (d' = z(H) - z(F)). Increase in d' signifies improved signal detection, i.e. a better outcome. A d' near zero indicates a performance at chance, i.e., a poor performance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 18 | 20
arbitrary units | 2.45 (0.95) | 2.34 (0.58) | 2.66 (0.93)

5. Primary Outcome: D-prime Score
Description: The Dot Pattern Expectancy (DPX) task is an adaptation of the expectancy AX task that uses pairs of simple dot patterns rather than letter pairs as stimuli. The DPX task will be performed in 3 blocks. Each trial consists of a cue dot pattern followed by a probe dot pattern. Different combinations of cues and probes enable the identification of a specific deficit in a subject's ability to maintain goal-relevant information throughout a trial. Timing will be jittered and each block of the DPX task will consist of 40 trials: 24 AX (60%), 6 AY (15%), 6 BX (15%) and 4 BY (10%). Each block will last 6 minutes. d'-context will be calculated as a measure of signal detection, which indicates the normalized rate of AX hits to BX false positives (d' = z(H) - z(F)). Increase in d' -context signified improved signal detection, i.e. a better outcome. A d' near zero indicates a performance at chance, i.e., a poor performance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 18 | 20
arbitrary units | 3.47 (0.88) | 3.36 (0.75) | 3.10 (0.91)

6. Primary Outcome: Changes in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: Intends to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. The composite score is reported as a T-score, with a mean of 50 and standard deviation of 10. Higher values indicate greater cognitive functioning.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 17 | 20
T-score | 53.3 (11.1) | 53.6 (6.01) | 54 (11.9)

7. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: as for outcome 1
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 16 | 10 | 17
arbitrary units | 23 (4.3) | 20.3 (2.8) | 23.8 (3.5)

8. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: as for outcome 1
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 9 | 15
arbitrary units | 23.1 (4.7) | 19.8 (4.0) | 24.2 (3.5)

9. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: as for outcome 2
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 16 | 9 | 17
z-score | -0.33 (0.51) | 0.09 (0.54) | -0.44 (0.44)

10. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: as for outcome 2
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 9 | 15
z-score | -0.24 (0.48) | -0.38 (0.42) | -0.4 (0.49)

11. Primary Outcome: D-prime Score
Description: as for outcome 4
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 16 | 10 | 17
arbitrary units | 3.24 (0.74) | 3.07 (0.52) | 3 (1.05)

12. Primary Outcome: D-prime Score
Description: as for outcome 4
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 10 | 15
arbitrary units | 3.22 (0.88) | 3.37 (0.75) | 3.18 (1.27)

13. Primary Outcome: Changes in DPX Task Performance
Description: as for outcome 5
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 16 | 10 | 17
arbitrary units | 2.90 (1.02) | 3.71 (0.45) | 2.84 (1.04)

14. Primary Outcome: Changes in DPX Task Performance
Description: as for outcome 5
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 10 | 15
arbitrary units | 2.92 (0.91) | 3.72 (0.81) | 2.91 (1.12)

15. Primary Outcome: Changes in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 6
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 17 | 10 | 18
T-score | 57.9 (9.9) | 57.8 (8.04) | 56.1 (10.8)

16. Primary Outcome: Changes in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 6
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 9 | 15
T-score | 59.1 (9.7) | 62.2 (6.22) | 60.2 (11.2)

17. Primary Outcome: Changes in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 6
Time Frame: follow up (week 24)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 9 | 15
T-score | 60.8 (6.6) | 61.1 (8.2) | 63.3 (8.1)

18. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: as for outcome 3
Time Frame: mid-test (week 6)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 10 | 17
z-score | -0.25 (0.42) | -0.09 (0.57) | -0.44 (0.29)

19. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: as for outcome 3
Time Frame: post-test (week 12)
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 10 | 15
z-score | -0.16 (0.52) | -0.25 (0.36) | -0.25 (0.24)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: assessed adverse events during the 12 weeks that individuals completed tDCS. They were asked after each session if they had an adverse reaction during the tDCS session.
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 2/20 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/18 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Active-tDCS (N=20) | Left Active-tDCS (N=18) | Sham tDCS (N=20)
Temporary moderate/severe tDCS headband discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT03896425/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03896425/ICF_001.pdf